CLINICAL TRIAL: NCT04183582
Title: A Two Phase Pilot of a Behavioural Activation (BA) Programme Specifically Adapted to Support Women Experiencing Postnatal Low Mood in Blackpool
Brief Title: Behavioural Activation (BA) for Postnatal Depression in Blackpool
Acronym: BA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Society for the Prevention of Cruelty to Children (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBS001
Record Dates: First submitted 2019-11-26; First posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Postnatal Depression
Keywords: Psychoeducation, Mental Health, Depression, Postnatal
MeSH Terms: conditions — Depression, Postpartum; Psychological Well-Being; Depression

STUDY DESIGN:
Intervention Model Description: Experimental Arm - single group study
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Single arm group receiving Behavioural Activation, a facilitated self-help programme delivered by trained Health Visitors as six one hour sessions over four weeks.
  Interventions: Behavioral: Behavioural Activation

INTERVENTIONS:
Behavioral: Behavioural Activation — Behavioural Activation is a treatment for depression, the current programme has been adapted to suit the needs of postnatal women Session 1: Getting Started Session 2: Identifying Triggers, Reactions and Avoidance Patterns (TRAPs) Session 3: Turning TRACs in to Triggers, Reactions and Alternative Coping (TRACs) Session 4: Support and Communication Session 5: Being a "Good Enough" Mum Session 6: Staying Well

SUMMARY:
Is Behavioural Activation feasible, acceptable and potentially effective for mothers experiencing post natal depression in Blackpool?

Phase 1: A series of single case studies which aim to examine and refine a) the appropriateness of the programme to women in Blackpool b) the suitability of BA as part of a stepped-care approach to perinatal mental health within the Health Visitor pathway and c) the delivery of the programme in practice.

Phase 2: A preliminary single group study examining the quantitative outcomes for participating women (i.e. symptoms of depression, anxiety and general mood, parental stress, responsiveness, and behavioural avoidance and activation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Score between 10-19 on PhQ9
* Have given birth within the last 6 months
* Willing to engage in a psychological therapy
* Informed, prepared and safe to participate in the programme
* Able to understand spoken and basic written English

Exclusion Criteria:

* Under 18 years old
* Score under 10 or over 19 on the PHQ9
* Receiving another from of psychological treatment for depression
* Unwilling to engage in a psychological therapy
* Another primary area of difficulty which takes precedence over the current programme (e.g.substance dependency disorders, suicidal crises, frequent, serious and deliberate self-harm, acute threat in the form of serious interpersonal violence from a partner or friend or family member, and evidence of more serious mental health disorders which may require additional support, i.e., psychotic disorders, Bipolar Disorder

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ9) | Baseline, 6 weeks, 18 weeks, 1 year
  The PHQ9 is a 9-item multi-purpose instrument which can be used to screen, diagnose, monitor and assess symptoms of depression.
Generalised Anxiety Disorder Questionnaire (GAD7) | Baseline and 6 weeks
  The GAD7 is a 7-item multi-purpose instrument which can be used to screen, diagnose, monitor and assess symptoms of anxiety.
Parental Stress Scale (PSS) | Baseline and 6 weeks
  The PSS is a self-report scale that intended to assess parental stress. It contains 18 items representing pleasure or positive themes of parenthood (emotional benefits, self-enrichment, personal development) and negative components (demands on resources, opportunity costs and restrictions).
Maternal Infant Responsiveness Instrument (MIRI) | Baseline and 6 weeks
  The MIRI is a 22-item scale designed to measure the parent's feelings about the infant and an appraisal of their infant's responsiveness.
Behavioural Activation for DEpression Scale (BADS) | Baseline and 6 weeks
  The BADS is a 25-item scale which can track change in behaviours which are hypothesised to underlie depression which are specifically targeted through Behavioural Activation. It comprises of four subscales; activation, avoidance/rumination, work/school impairment and social impairment.
Snaith-Hamilton Pleasure Scale (SHAPS) | Baseline and 6 weeks
  The SHAPS is a 14-item measure of anhedonia (the degree to which an individual is able to experience pleasure). It comprises of four subscales which measure response/hedonic experiences; interests/past-times, social interaction, sensory experiences, food/drink.

SECONDARY OUTCOMES:
Ages and Stages Questionnaire (ASQ) | Data collected when child is 1 year and 2-2.5years
  Nationally mandated data collected by Health Visitors in the UK to assess children's development. This includes five key areas of development, communication, gross motor, fine motor, problem solving, and personal-social.

OTHER OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) | Baseline, 2 week (x2), 3 weeks (x2), 4 weeks, 5 weeks, 6 weeks
  The EPDS is a 10-item measure which assesses low mood and symptoms of depression. It has been designed specifically for women in the postnatal period.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Early Child Development, Blackpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No
To be confirmed with programme developers, research team and potential academic partners